CLINICAL TRIAL: NCT06696898
Title: Effects of Somatosensory Motor Control With and Without Myofascial Release on Pain, Lumbar Range of Motion and Functional Disability in Patients With Sciatica
Brief Title: Effects of SSMC With and Without Myofascial Release in Patients With Sciatica
Acronym: Sciatica
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0238
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sciatica Pain; Sciatica
Keywords: Sensorimotor Training; PNF Exercises; Functional Disability
MeSH Terms: conditions — Sciatica | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatosensory Motor Control & Myofascial Release (Experimental): A series of proprioceptive and neuromuscular control exercises targeting lumbar stability and pain reduction.Somatosensory Motor Control & Myofascial Release Procedure.MFR is Manual therapy technique that focused on releasing fascial restrictions to improve lumbar mobility and decrease pain.
  Interventions: Procedure: Somatosensory Motor Control Exercises; Procedure: Myofascial Release Technique
- Sensorimotor training (Active Comparator): Somatosensory motor control are Structured exercises aimed at enhancing proprioception and motor control to reduce pain and improve function in sciatica patients.
  Interventions: Procedure: Sensorymotor training

INTERVENTIONS:
Procedure: Somatosensory Motor Control Exercises — The Somatosensory motor control training protocol assembled into three components, 1) PNF exercises (Each patient alternately contracted trunk extensors and flexors isometrically for 10 seconds against maximum resistance while seated, then contracted trunk agonists alternately in a concentric and eccentric manner against manual resistance without relaxing, then moved his or her trunk in a twisting and diagonal orientation against maximum resistance), 2) Somatosensory exercises in which a wobbling board was used and six types of exercises were performed including hallowing, one lower limb elevation, opposite upper and lower limb elevation from a four-limb supported position (quadruped), abdominal reinforcement, maintaining a bridging posture, and one lower limb elevation from the bridging posture, and 3) finally Vestibular training which involved exercises to improve gaze focus, exercises for enhancing eye movements.
  Arms: Somatosensory Motor Control & Myofascial Release
Procedure: Myofascial Release Technique — Manual therapy technique that applies sustained pressure to myofascial tissues around the lumbar spine and pelvis to release tension and improve mobility.Myofascial Release Technique MFR is given with the ulnar border from proximal to distal direction with a light gentle pressure over the hamstring muscle until the slack in the skin is loosened. (2) Every strike is to be held for 30 seconds, 5 repetitions per session
  Arms: Somatosensory Motor Control & Myofascial Release
Procedure: Sensorymotor training — The Somatosensory motor control training protocol assembled into three components, 1) PNF exercises (Each patient alternately contracted trunk extensors and flexors isometrically for 10 seconds against maximum resistance while seated, then contracted trunk agonists alternately in a concentric and eccentric manner against manual resistance without relaxing, then moved his or her trunk in a twisting and diagonal orientation against maximum resistance), 2) Somatosensory exercises in which a wobbling board was used and six types of exercises were performed including hallowing, one lower limb elevation, opposite upper and lower limb elevation from a four-limb supported position (quadruped), abdominal reinforcement, maintaining a bridging posture, and one lower limb elevation from the bridging posture, and 3) finally Vestibular training which involved exercises to improve gaze focus, exercises for enhancing eye movements.
  Arms: Sensorimotor training

SUMMARY:
Sciatica involves a radiating pain along the sciatic nerve, extending from the lower back through the hips and buttocks to each leg. Typically resulting from a herniated disk or spinal stenosis, this condition causes nerve compression that leads to pain, inflammation, and often numbness in the affected leg. Studies have shown that sensorimotor training with myofascial release can be effective in improving pain, lumbar range of motion and functional disability. The aim of this study is to evaluate the effects of Sensorimotor control training with and without myofascial releases on Pain, Lumbar range of motion and functional disability due to sciatica. Participants which meet inclusion criteria will be randomly allocated using online randomization tool into two groups. Group A will receive somatosensory control training with Routine Physical Therapy for 45 minutes with short resting interval for Group B will receive Somatosensory training with myofascial release technique for 45min. Each group will receive treatment sessions of 3 days per week for 12 weeks.

DETAILED DESCRIPTION:
Despite the considerable body of research addressing sciatica and various therapeutic interventions, there remains a significant gap in understanding the comparative effectiveness of combining somatosensory motor control exercises with myofascial release techniques specifically for this condition.

The role of somatosensory motor control in managing sciatica has gained considerable attention in the last decade.The author conducted research on neural mobilization and somatosensory motor control training on individual with persistent low back pain (2023). They involved forty-five individuals that have been classified into three groups and applying different treatment strategies on study groups. Neural mobilization and somatosensory training are effective in relief of pain and improve lumbar range of motion. They concluded that adding the neural mobilization and somatosensory training to routine physical therapy were equally effective on sciattica. The other author stated that patients with sciatica often exhibit impaired motor control, which contributes to pain and functional limitations. Their study suggested that targeted exercises to improve somatosensory motor control could alleviate symptoms and enhance lumbar function. This finding has been supported by subsequent studies, which emphasized the importance of neuromuscular re-education in sciatica management. The research was conducted by Faraz et al. (2024) to check the effectiveness of myofascial release technique on range of motion and functional disability for patients with piriformis syndrome. They include sixty-six participants with deep gluteal syndrome. They showed that between group analysis showed MFR technique along with conventional therapy was more effective in alleviating pain and functional disability as compared to routine physical therapy .

This study aims to fill this gap by investigating the combined effects of somatosensory motor control and myofascial release on pain reduction, lumbar range of motion, and functional disability in sciatica patients. Most studies have focused either on general low back pain or on single interventions without evaluating the synergistic effects of comprehensive treatment protocols. Furthermore, limited research exists on the implementation of these combined therapies within the Pakistani population, where cultural, socioeconomic, and healthcare access factors may influence treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient Diagnosed with sciatica (confirmed by clinical examination and imaging)
* Patient with Unilateral sciatica pain
* Patient Experiencing symptoms for at least 3 months
* Pain (VAS) score ≥ 5) in the lumbar and/or lower extremity region in patients.
* The disability with a score of at least 20% by the Oswestry Disability Index (
* Stable patient , no recent changes in treatment regimen for sciatica within the past 4 weeks

Exclusion Criteria:

* Patients with Lumbar spine surgery history within the past 6 months (11)
* Patients who have been Another clinical trial participant within the past 3 months (1).
* Patients with Physical therapy interventions contraindicated like in Severe cardiovascular disease and Uncontrolled hypertension Acute disc herniation requiring urgent surgical intervention (10).
* Patients with Significant comorbidities like malignancy, spinal infection and Severe osteoporosis affecting spine stability (14).
* Inability in patients to communicate effectively in Urdu or English, hindering comprehension of study instructions and assessments.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) (For functional disability) | 4th week
  There are Total 10 Questions and each question, there is a possible 5 points: 0 for the first answer, 1 for the second answer, etc. Add up the total for the 10 questions and rate them on the scale at right. The ODI has good internal consistency (Cronbach α .86) and test-retest reliability (0.84). The scoring Interpretations of Oswestry Disability Index is 0% to 20%: minimal disability, 21-40% moderate disability, 41-60% severe Disability, 61-80% crippled and 81-100% are bed bound or exaggerating their symptoms.
Visual Analog Scale (For Pain) | 1st day
  The VAS is a horizontal or vertical line, usually 10 centimeters (100 mm) in length. The ends are defined as the extreme limits of pain (e.g., "no pain" to "worst pain imaginable"). The participant is asked to mark on the line the point that represents their perception of their current pain level. A score 0mm No Pain, 30mm Mild Pain, 50mm Moderate Pain, 70mm severe Pain and 100mm Worst Pain imaginable
Modified Schober Test:(For Lumbar range of motion) | 4th week
  In this Ask the participant to stand upright with feet together and mark a point 10 cm below and 5 cm above the L5 spinous process (the dimples of Venus and 10 cm caudally) and calculated by Subtract the baseline measurement (S1) from the flexion measurement (S2) to calculate the range of lumbar spine flexion. The difference between S1 and S2 represents the lumbar spine flexion range in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Phd, Principal Investigator — Riphah International University
Locations (1):
- Well Versed Physio clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostelo RW. Physiotherapy management of sciatica. J Physiother. 2020 Apr;66(2):83-88. doi: 10.1016/j.jphys.2020.03.005. Epub 2020 Apr 11. No abstract available. PMID 32291226
- [Background] Fairag M, Kurdi R, Alkathiry A, Alghamdi N, Alshehri R, Alturkistany FO, Almutairi A, Mansory M, Alhamed M, Alzahrani A, Alhazmi A. Risk Factors, Prevention, and Primary and Secondary Management of Sciatica: An Updated Overview. Cureus. 2022 Nov 12;14(11):e31405. doi: 10.7759/cureus.31405. eCollection 2022 Nov. PMID 36514653
- [Background] Bello B, Danazumi MS, Kaka B. Comparative Effectiveness of 2 Manual Therapy Techniques in the Management of Lumbar Radiculopathy: A Randomized Clinical Trial. J Chiropr Med. 2019 Dec;18(4):253-260. doi: 10.1016/j.jcm.2019.10.006. Epub 2020 Sep 3. PMID 32952470
- [Background] Brumagne S, Diers M, Danneels L, Moseley GL, Hodges PW. Neuroplasticity of Sensorimotor Control in Low Back Pain. J Orthop Sports Phys Ther. 2019 Jun;49(6):402-414. doi: 10.2519/jospt.2019.8489. PMID 31151373
- [Background] Khan T, Rizvi MR, Sharma A, Ahmad F, Hasan S, Uddin S, Sidiq M, Ammari A, Iqbal A, Alghadir AH. Assessing muscle energy technique and foam roller self-myofascial release for low back pain management in two-wheeler riders. Sci Rep. 2024 May 27;14(1):12144. doi: 10.1038/s41598-024-62881-8. PMID 38802553
- [Background] Ozsoy G, Ilcin N, Ozsoy I, Gurpinar B, Buyukturan O, Buyukturan B, Kararti C, Sas S. The Effects Of Myofascial Release Technique Combined With Core Stabilization Exercise In Elderly With Non-Specific Low Back Pain: A Randomized Controlled, Single-Blind Study. Clin Interv Aging. 2019 Oct 9;14:1729-1740. doi: 10.2147/CIA.S223905. eCollection 2019. PMID 31631992
- [Background] Ozog P, Weber-Rajek M, Radziminska A, Goch A. Analysis of Postural Stability Following the Application of Myofascial Release Techniques for Low Back Pain-A Randomized-Controlled Trial. Int J Environ Res Public Health. 2023 Jan 26;20(3):2198. doi: 10.3390/ijerph20032198. PMID 36767565
- [Background] van Dieen JH, Reeves NP, Kawchuk G, van Dillen LR, Hodges PW. Motor Control Changes in Low Back Pain: Divergence in Presentations and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):370-379. doi: 10.2519/jospt.2019.7917. Epub 2018 Jun 12. PMID 29895230
- [Background] Goossens N, Janssens L, Brumagne S. Changes in the Organization of the Secondary Somatosensory Cortex While Processing Lumbar Proprioception and the Relationship With Sensorimotor Control in Low Back Pain. Clin J Pain. 2019 May;35(5):394-406. doi: 10.1097/AJP.0000000000000692. PMID 30730445
- [Background] Marchand F, Laudner K, Delank KS, Schwesig R, Steinmetz A. Effects of Sensorimotor Training on Transversus Abdominis Activation in Chronic Low Back Pain Patients. J Pers Med. 2023 May 11;13(5):817. doi: 10.3390/jpm13050817. PMID 37240987
- [Background] Amjad F, Mohseni-Bandpei MA, Gilani SA, Ahmad A, Waqas M, Hanif A. Urdu version of Oswestry disability index; a reliability and validity study. BMC Musculoskelet Disord. 2021 Mar 29;22(1):311. doi: 10.1186/s12891-021-04173-0. PMID 33781267
- [Background] Jenks A, Hoekstra T, van Tulder M, Ostelo RW, Rubinstein SM, Chiarotto A. Roland-Morris Disability Questionnaire, Oswestry Disability Index, and Quebec Back Pain Disability Scale: Which Has Superior Measurement Properties in Older Adults With Low Back Pain? J Orthop Sports Phys Ther. 2022 Jul;52(7):457-469. doi: 10.2519/jospt.2022.10802. Epub 2022 May 18. PMID 35584027
- [Background] Xu HR, Zhang YH, Zheng YL. The effect and mechanism of motor control exercise on low back pain: a narrative review. EFORT Open Rev. 2023 Jul 3;8(7):581-591. doi: 10.1530/EOR-23-0057. PMID 37395680
- [Background] Tousignant M, Poulin L, Marchand S, Viau A, Place C. The Modified-Modified Schober Test for range of motion assessment of lumbar flexion in patients with low back pain: a study of criterion validity, intra- and inter-rater reliability and minimum metrically detectable change. Disabil Rehabil. 2005 May 20;27(10):553-9. doi: 10.1080/09638280400018411. PMID 16019864